CLINICAL TRIAL: NCT06980389
Title: Node-Sparing Short-Course Radiotherapy Followed by First-Line Therapy Plus PD-1 Inhibitor in Unresectable Locally Advanced or Metastatic pMMR/MSS Gastric Cancer: A Prospective, Randomized, Controlled Phase II Trial (MODIFI-GC)
Brief Title: Node-Sparing Short-Course Radiotherapy Plus First-Line Therapy and PD-1 Inhibitor in Unresectable/Metastastic pMMR/MSS Gastric Cancer (MODIFI-GC)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanxin Luo,MD, MD, PhD, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZSLYEC-226
Record Dates: First submitted 2025-04-24; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Immune Checkpoint Therapy; Radiotherapy; Metastatic Gastric Carcinoma
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Node-sparing Radiotherapy Group (Experimental)
  Interventions: Combination Product: Node-Sparing Radiotherapy plus first-line therapy
- First-line therapy Group (Active Comparator)
  Interventions: Combination Product: First-line treatment

INTERVENTIONS:
Combination Product: Node-Sparing Radiotherapy plus first-line therapy — Patients will receive node-sparing modified short-course radiotherapy, followed by standard first-line chemotherapy combined with a PD-1 inhibitor starting 2-5 days after radiotherapy. Treatment will continue until disease progression or the occurrence of unacceptable toxicity.
  Arms: Node-sparing Radiotherapy Group
Combination Product: First-line treatment — Patients will receive standard first-line chemotherapy combined with a PD-1 inhibitor. Treatment will continue until disease progression or the occurrence of unacceptable toxicity.
  Arms: First-line therapy Group

SUMMARY:
For patients with unresectable locally advanced or metastatic gastric cancer, systemic anti-tumor therapy remains the mainstay of treatment. Combining chemotherapy with immune checkpoint inhibitors has gradually become the standard first-line treatment for advanced gastric cancer. Radiotherapy can enhance the release of tumor-associated antigens, thereby improving the responsiveness of MSS/pMMR tumors to PD-1 inhibitors. Tumor-draining lymph nodes (TDLNs) are key sites for the anti-tumor activity of PD-1 blockade; however, radiation-induced damage and fibrosis may impair lymphatic drainage and local immune responses. Previous studies have suggested that irradiation of the primary tumor combined with immune checkpoint blockade can produce an abscopal effect, mediating regression of distant metastases. This study aims to evaluate whether node-sparing modified short-course radiotherapy followed by chemotherapy and PD-1 blockade can improve 2-year progression-free survival (PFS) in patients with unresectable locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signs a written informed consent form.

  * Aged between 18 and 75 years at the time of enrollment.
  * Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
  * Expected survival of more than 3 months.
  * At least one measurable lesion as defined by RECIST 1.1.
  * Histologically confirmed unresectable locally advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction.
  * Tumor biopsy indicates proficient mismatch repair (pMMR) based on positive immunohistochemical staining for MSH1, MSH2, MSH6, and PMS2, or microsatellite stability (MSS) by genetic testing.
  * No prior systemic anti-tumor therapy before study treatment, including radiotherapy, chemotherapy, immunotherapy, biologics, or small-molecule targeted therapy.
  * Agrees to provide tumor tissue and peripheral blood samples during screening and throughout the study for research purposes.
  * Adequate organ function as defined below:
  * Hematologic (without blood transfusion or hematopoietic growth factor support within 7 days prior to treatment):
  * Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L
  * Platelet count ≥ 100 × 10⁹/L
  * Hemoglobin ≥ 90 g/L
  * Renal:
  * Calculated creatinine clearance (CrCl) ≥ 50 mL/min using the Cockcroft-Gault formula:

CrCl = [(140 - age) × weight (kg) × 0.85 (if female)] / [72 × serum creatinine (mg/dL)]

* Urine protein < 2+ by dipstick or < 1.0 g/24 h
* Hepatic:
* Total bilirubin (TBil) ≤ 1.5 × upper limit of normal (ULN)
* AST and ALT ≤ 2.5 × ULN
* Serum albumin ≥ 28 g/L
* Coagulation:
* INR and APTT ≤ 1.5 × ULN
* Cardiac:
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Women of childbearing potential must have a negative urine or serum pregnancy test within 3 days prior to study treatment. If urine test is inconclusive, a serum test result shall prevail. Women of childbearing potential who are sexually active with non-sterilized male partners must agree to use an acceptable method of contraception from screening through 120 days after the last dose of study drug. Whether to discontinue contraception after this period should be discussed with the investigator. Periodic abstinence and calendar methods are not acceptable.
* Women of childbearing potential are defined as those who have not undergone surgical sterilization (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) and who are not postmenopausal (defined as ≥12 months of amenorrhea without alternative medical cause and with serum FSH levels in the postmenopausal range).
* Highly effective contraception methods are those with a failure rate <1% per year when used consistently and correctly. In addition to barrier methods, hormonal contraception (e.g., oral contraceptives) must also be used.
* Willing and able to comply with all scheduled visits, treatment plans, laboratory tests, and other study requirements.

Exclusion Criteria:

* • Radiotherapy within 4 weeks prior to enrollment or radionuclide therapy within 8 weeks, except for palliative radiotherapy to bone metastases.

  * History of other malignancies within 5 years prior to enrollment, except for those considered cured by local therapy, such as basal cell carcinoma, squamous cell carcinoma of the skin, superficial bladder cancer, or ductal carcinoma in situ of the breast.
  * Gastrointestinal perforation and/or fistula within 6 months prior to enrollment.
  * Clinically significant bowel obstruction.
  * Symptomatic central nervous system (CNS) metastases.
  * Diagnosis of HER2-positive gastric or gastroesophageal junction adenocarcinoma.
  * Inability to swallow oral medications, malabsorption syndrome, or any other condition affecting gastrointestinal absorption.
  * Prior systemic or local anti-tumor therapy for gastric cancer, including curative surgery, chemotherapy, radiotherapy, immunotherapy (e.g., immune checkpoint inhibitors, agonists, or cell therapy), biologics, or small-molecule targeted agents.
  * Receipt of nonspecific immunomodulatory agents (e.g., interleukins, interferons, thymic peptides, tumor necrosis factor) within 2 weeks prior to study treatment (excluding IL-11 for thrombocytopenia); use of anti-tumor traditional Chinese medicine within 1 week prior to study treatment.
  * Active autoimmune disease requiring systemic therapy within the past 2 years (e.g., corticosteroids, immunosuppressants, DMARDs). Replacement therapy (e.g., thyroid hormone, insulin, or physiologic corticosteroids for adrenal/pituitary insufficiency) is permitted.
  * History of or current interstitial lung disease or non-infectious pneumonitis requiring systemic corticosteroids.
  * History of significant bleeding disorders or coagulopathy; current or prior long-term anticoagulation (e.g., atrial fibrillation with CHADS2 score ≥ 2).
  * Uncontrolled comorbidities including, but not limited to, decompensated cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe active peptic ulcer or gastritis, or psychiatric/social conditions interfering with protocol compliance or informed consent.
  * History of myocarditis, cardiomyopathy, or malignant arrhythmia; unstable angina, heart failure requiring hospitalization, or vascular disease (e.g., aortic aneurysm requiring repair or DVT) within 12 months before treatment; other cardiac conditions that may interfere with safety evaluation, such as poorly controlled arrhythmias, myocardial infarction, or ischemia.
  * Within 6 months prior to treatment: gastroesophageal varices, severe ulcers, unhealed wounds, GI perforation, fistula, intestinal obstruction, intra-abdominal abscess, or acute GI bleeding.
  * Arterial thromboembolism, grade ≥3 venous thromboembolism (per NCI CTCAE v5.0), TIA, stroke, hypertensive crisis, or hypertensive encephalopathy within 6 months before treatment.
  * Acute exacerbation of COPD within 1 month prior to treatment; uncontrolled hypertension (SBP ≥ 160 mmHg or DBP ≥ 100 mmHg despite oral therapy).
  * Active or prior history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis) or chronic diarrhea.
  * Serious infection within 4 weeks prior to treatment, including those requiring hospitalization, sepsis, or severe pneumonia; active systemic infection requiring anti-infective therapy within 10 days before treatment (excluding antiviral therapy for HBV or HCV).
  * Major surgery or significant trauma within 30 days prior to treatment; minor local surgery within 3 days prior (excluding central venous catheter placement via peripheral vein).
  * History of immunodeficiency; HIV antibody positive; long-term use of systemic corticosteroids or immunosuppressants.
  * Known active tuberculosis (TB), or suspected active TB not ruled out by clinical assessment (e.g., sputum testing, chest imaging); known active syphilis.
  * History of allogeneic organ or hematopoietic stem cell transplantation.
  * Untreated active hepatitis B infection (HBsAg positive and HBV DNA > 1,000 copies/mL or 200 IU/mL); patients with HBV must receive antiviral therapy during the study. Active hepatitis C infection (HCV antibody positive with detectable HCV RNA) is also excluded.
  * Receipt of a live vaccine within 30 days prior to treatment or planned during the study period.
  * Known allergy to any component of study drugs or history of severe hypersensitivity to monoclonal antibodies.
  * Known history of psychiatric disorders, substance abuse, alcoholism, or drug addiction.
  * Pregnant or breastfeeding women.
  * Any condition, treatment, or abnormal laboratory findings that may confound study results, interfere with study participation, or not be in the best interest of the participant.
  * Local or systemic disease caused by benign tumors, or tumor-related complications with high medical risk or uncertain prognosis (e.g., leukemoid reaction with WBC > 20 × 10⁹/L, cachexia with >10% weight loss in 3 months before screening, or BMI ≤ 18).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-05-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From initiation of treatment until disease progression or death, whichever occurs first, assessed over a period of up to 24 months

SECONDARY OUTCOMES:
Objective response rate | From the start of treatment until disease progression, assessed over a period of up to 24 months
Duration of response | From the first documented occurrence of complete response (CR) or partial response (PR) to the first documented disease progression (per RECIST v1.1) or death from any cause, whichever occurs first, assessed over a period of up to 24 months
Disease control rate | From treatment start to the end of study at 2 years
Overall survival (OS) rate | From treatment start to the end of study at 2 years
Treatment related adverse effect | From treatment start to 30 days after the end of treatment
R0 resection rate | From treatment start to the end of study at 2 years
Quality of life by EORTC QLQ-C30 | From treatment start to the end of study at 2 years
EORTC QLQ-STO22 | From treatment start to the end of study at 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No